CLINICAL TRIAL: NCT07114172
Title: Study of Melanoma-Resistant PET Monitoring Based on Key Rate-limiting Enzymes for Fatty Acid Metabolism in Healthy Volunteers
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: KY20252266
Record Dates: First submitted 2025-08-04; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-07

CONDITIONS: Melanoma (Skin Cancer); Health Volunteers; PET / CT
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Safety assessment (Experimental)
  Interventions: Diagnostic Test: 68Ga-ACC-DE/68Ga-FASN-DE/68Ga-ACLY-DE PET/CT

INTERVENTIONS:
Diagnostic Test: 68Ga-ACC-DE/68Ga-FASN-DE/68Ga-ACLY-DE PET/CT — Recruit 15 healthy adult volunteers, divided into three groups, to undergo dynamic PET/CT (1 hour) and static PET/CT (2 hours and 3 hours) imaging with 68Ga-ACC-DE, 68Ga-FASN-DE, or 68Ga-ACLY-DE, respectively, to assess safety, biodistribution, and radiation dosimetry, laying the foundation for subsequent studies.

SUMMARY:
This is a small-sample safety study involving 15 healthy volunteers who were divided into groups and underwent 68Ga-ACC-DE, 68Ga-FASN-DE, and 68Ga-ACLY-DE PET/CT imaging for safety, biodistribution, and radiation dosimetry assessments, laying the foundation for subsequent studies on the efficacy of resistance monitoring in melanoma targeted therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 to 65 years old (including the boundary values); Gender: Male or female; Weight: Male weight ≥ 50 kg, female weight ≥ 45 kg, and body mass index (BMI = weight (kg) / height² (m²)) within the range of 18.0 to 28.0 kg/m² (including boundary values); Participants must fully understand and voluntarily participate in this experiment and sign an informed consent form.

Exclusion Criteria:

* Individuals who cannot tolerate intravenous administration (e.g., those with a history of fainting from needles or blood); Individuals with alcohol allergies; Pregnant or breastfeeding women; Individuals with severe diseases of the heart, kidneys, lungs, blood vessels, nervous system, or mental health, immune deficiency diseases, or hepatitis/cirrhosis; Individuals whom the investigator deems unsuitable for or unable to complete PET or other imaging examinations for special reasons; Other circumstances deemed by the investigator to be unsuitable for participation in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-08-15 (Estimated); Primary Completion 2025-10-15 (Estimated); Study Completion 2025-10-15 (Estimated)

PRIMARY OUTCOMES:
The maximum standardized uptake value (SUVmax) | One hour after injection of the tracer
  The maximum standardized uptake value (SUVmax) of 68Ga-ACC-DE/68Ga-FASN-DE/68Ga-ACLY-DE in the target population.

IPD SHARING:
Plan to Share IPD: No